CLINICAL TRIAL: NCT02897193
Title: 3.2 mm Diameter Implants and Soft Tissue Grafts in Alternative to Horizontal Bone Augmentation for Placing 4.2 mm Diameter Implants at Central Incisors. A Multicenter Randomised Controlled Trial
Brief Title: Central Incisors Narrow Implants in Alternative to Bone Augmentation With 4.2 mm Implants .
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Alpha - Bio Tec Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABT-ME-130815
Record Dates: First submitted 2016-09-01; First posted 2016-09-13 (Estimated); Last update posted 2019-07-16 (Actual); Status verified 2019-06

CONDITIONS: Upper Central Incisor Edentulism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dental implant with bone augmentation (Active Comparator): patients will be installed with ICE Dental implant 4.2 mm diameter with Alpha-Bio's grafts horizontal bone augmentation
  Interventions: Device: ICE dental implant 4.2 mm; Device: Alpha Bio's Graft Bovine bone; Device: Alpha Bio's Graft resorbable membrane
- narrow implant (Experimental): patients will be installed with NICE Dental implant 3.2 mm diameter
  Interventions: Device: NICE dental implant 3.2 mm

INTERVENTIONS:
Device: ICE dental implant 4.2 mm — ICE dental implant 4.2 mm diameter
  Arms: Dental implant with bone augmentation
Device: NICE dental implant 3.2 mm — NICE dental implant 4.2 mm diameter
  Arms: narrow implant
Device: Alpha Bio's Graft Bovine bone — Alpha Bio's Graft Bovine Bone
  Arms: Dental implant with bone augmentation
Device: Alpha Bio's Graft resorbable membrane — Alpha Bio's Graft resorbable collagen membrane
  Arms: Dental implant with bone augmentation

SUMMARY:
Horizontal bone augmentation procedures are commonly used to increase bone width to allow the placement of dental implants or to improve aesthetics in deficient areas. Smaller diameter implants could be used instead in order to avoid bone augmentation procedures.

The comparison between these two solutions will be evaluated in the trial.

ELIGIBILITY:
Inclusion Criteria:

* Upper central incisor edentulism
* bone width between 3.5-4.5 mm
* requirement of only one implant supported crown
* patient is willing to sign an informed consent

Exclusion Criteria:

* General contraindications to implant surgery.
* Immunosuppressed or immunocompromised patients
* Patients irradiated in the head and neck area.
* Patients with poor oral hygiene and motivation.
* Uncontrolled diabetes.
* Pregnancy or lactation.
* Addiction to alcohol or drugs.
* Untreated periodontal disease.
* Treated or under treatment with intravenous amino-biphosphonates.
* Poor oral hygiene and motivation.
* Psychiatric problems and/or unrealistic expectations.
* Acute infection (abscess) or suppuration in the area intended for implant placement.
* Patients referred only for implant placement if cannot be followed at the treatment centre.
* Patient unable to attend the follow-up controls for 3 years after implant loading.
* Patient included in other studies, if this protocol cannot be properly followed.
* Immediate post-extractive sites (to be eligible at least 3 months must have passed since extraction).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-08; Primary Completion 2019-09 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
bone loss | 2 years
  bone loss level as will be measured from the radio-graphic images

SECONDARY OUTCOMES:
Cumulative implant survival | 2 years
  Counting number of survived implants at the end of the study

CONTACTS AND LOCATIONS:
Locations (2):
- Chile (2):
  - University of Antofagasta, Antofagasta
  - Andrés Bello National University, Santiago

REFERENCES:
- See also: sponsor site — http://www.alpha-bio.net